CLINICAL TRIAL: NCT06804655
Title: Pharmacoscopy for Patients With Refractory Primary Brain Tumors
Acronym: EViDENCE-BT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other); University Hospital, Basel, Switzerland (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EViDENCE-BT
Record Dates: First submitted 2024-12-17; First posted 2025-02-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Brain (Nervous System) Cancers; Glioblastoma; Glioma; Ependymoma; Medulloblastoma; Meningioma; Rare Primary Brain Tumors; Rare CNS Primary Tumors
Keywords: pharmacoscopy; drug testing; refractory tumor; drug repurposing; personalized medicine
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms; Glioblastoma; Glioma; Ependymoma; Medulloblastoma; Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients will have their tumor analyzed by pharmacoscopy. (Experimental): Therapeutic decisions will be taken considering the results of the pharmacoscopy analysis, and also standard histopathological and molecular analysis, including next generation sequencing, molecular profiling analysis as available, characteristics of the patient and previous treatments received.
  Interventions: Device: Pharmacoscopy 1.0

INTERVENTIONS:
Device: Pharmacoscopy 1.0 — The intervention is the submission of freshly obtained surgical material to ex vivo drug profiling which we term pharmacoscopy (PCY). The performance study is interventional as the test results shall influence patient management decisions and/or may be used to guide treatment.

SUMMARY:
Advanced technology of ex vivo drug profiling referred to as pharmacoscopy may allow to identify novel drugs for the treatment of glioblastoma and other refractory brain tumors at an individual patient level. This personalized therapeutic approach was developed and validated in pre-clinical glioma models. With the current research proposal, we seek to establish feasibility for a clinical interventional trial for patients with refractory primary brain tumors that is based on pharmacoscopy-guided selection of treatment.

The study is supported by an unrestricted grant from Anti Cancer Fund.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older on day of signing informed consent, female or male.
2. Refractory glioblastoma, isocitrate dehydrogenase (IDH)-mutant astrocytoma or oligodendroglioma, histone-mutant glioma, ependymoma, medulloblastoma, meningioma or other rare primary brain tumor with a histological confirmation according to the WHO classification 2021. Primary tumors can be located at the cerebral or spinal level. Primary brain tumors with metastases outside of the brain may also be considered.
3. Karnofsky performance status of 60 or more
4. Life expectancy >12 weeks.
5. Limited systemic therapeutic options as per treating physician judgement. The number of previous lines of therapies is not limited.
6. Surgery clinically indicated. A histological confirmation of the diagnosis of a recurrent brain tumor will be required before any treatment can be initiated.
7. Adequate bone marrow, renal and hepatic function
8. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
9. Written informed consent for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Exclusion Criteria:

1. Inability to undergo brain or spine MRI.
2. Concurrent treatment with other systemic tumor-directed pharmacotherapies.
3. Intent to be treated with radiotherapy.
4. Any investigational antitumor therapy other than those under investigation in this study.
5. Judgment by the investigator that the patient should not participate in the study because the patient is unlikely to comply with study procedures, restrictions and requirements.
6. Intention to become pregnant during the course of the study or pregnancy. Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test.
7. Women who are breast feeding and who do not agree to discontinue nursing prior to the first study treatment and for the period defined in the protocol.
8. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the overall feasibility of pharmacoscopy-guided treatment for patients with refractory primary brain tumors | 2 months
  The feasibility is defined as:
  80% success rate of generating a pharmacoscopy result within 10 days of surgery (32/40 patients), 50% success rate of placing patients on selected drug based on pharmacoscopy (16/32 patients).

SECONDARY OUTCOMES:
To explore the efficacy of pharmacoscopy-guided treatment - 1 | 12 months
  (1) Response rate
To explore the efficacy of pharmacoscopy guided treatment - 2 | 12 months
  duration of response
To explore the efficacy of pharmascopy guided treatment - 3 | 12 months
  progression-free survival
To explore the efficacy of pharmascopy guided treatment - 4 | 24 months
  overall survival
To confirm the safety and tolerability of treatment selected based on pharmacoscopy - 1 | 12 months
  Neurological function (NANO scale, Nayak et al. 2017)
To confirm the safety and tolerability of treatment selected based on pharmacoscopy -2 | 12 months
  Karnofsky performance status (score 0-100)
To confirm the safety and tolerability of treatment selected based on pharmacoscopy - 3 | 12 months
  Steroid use (dose in mg equivalent dexamethasone)
Quality of life -1 | 12 months
  EORTC QLQ C30 auto-questionnaire
Quality of life - 2 | 12 months
  EORTC BN20 autoquestionnaire

OTHER OUTCOMES:
Translational research | 12 months
  prospective assessement of the value of liquid biopsy in parallel of imaging assessment

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel, Basel-Landschaft
  - Cantonal Hospital St Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Weiss T, Buhler M, Mena J, Lottenbach Z, Wegmann R, Sun M, Bihl M, Augustynek B, Baumann SP, Goetze S, van Drogen A, Pedrioli PGA, Penton D, Festl Y, Buck A, Kirschenbaum D, Zeitlberger AM, Neidert MC, Vasella F, Rushing EJ, Wollscheid B, Hediger MA, Weller M, Snijder B. High-throughput identification of repurposable neuroactive drugs with potent anti-glioblastoma activity. Nat Med. 2024 Nov;30(11):3196-3208. doi: 10.1038/s41591-024-03224-y. Epub 2024 Sep 20. PMID 39304781